CLINICAL TRIAL: NCT00595023
Title: GeneSearch Breast Lymph Node (BLN) Assay Timing Study
Status: Terminated | Type: Observational
Why Stopped: GeneSearch™ BLN Assay has been voluntarily withdrawn from the US market.
Sponsor: Janssen Diagnostics, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: GeneSearch BLN Timing Study; BLN-TIMING-2007.00
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Breast Cancer
Keywords: Sentinel lymph node; Metastasis
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Biological Assay

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: All eligible subjects
  Interventions: Device: GeneSearch™ Breast Lymph Node (BLN) Assay

INTERVENTIONS:
Device: GeneSearch™ Breast Lymph Node (BLN) Assay — The GeneSearch™ BLN Assay is a real time Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR) assay that detects the presence of breast tumor cell metastasis in lymph nodes through the detection of gene expression markers present in breast tissue, but not in nodal tissue (cell type specific messenger RNA).
  Other Names: BLN Assay; GeneSearch™ BLN Assay

SUMMARY:
This study is designed to collect data about the amount of time required to use the assay in clinical-use conditions.

DETAILED DESCRIPTION:
Assay turn-around-time will be collected at sites that are using the GeneSearch BLN Assay for intraoperative testing of sentinel lymph nodes. The sites must be planning to use the assay result to guide the decision to complete an axillary lymph node dissection.

ELIGIBILITY:
Inclusion Criteria:

* Pre-operatively established diagnosis of invasive carcinoma of the breast
* Scheduled for axillary sentinel lymph node dissection as per standard of care at the clinical site for newly diagnosed breast cancer patients
* Patients for whom the GeneSearch™ BLN Assay will be used intra-operatively to make a decision for an axillary lymph node dissection
* 18 years of age or older
* Female or male

Exclusion Criteria:

* Previous diagnosis of lymphoma
* Subjects participating in other research studies that would interfere with their full participation in this study
* Patients and/or conditions with 'interfering substances' as listed in the IFU
* Patients who have had any pre-operative treatment for breast cancer including neoadjuvant and/or hormonal intervention such as aromatase inhibitors or tamoxifen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intraoperative use of the GeneSearch™ BLN Assay to make a decision for an axillary lymph node dissection in patients with invasive carcinoma of the breast.
Sampling Method: Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To determine, under clinical use conditions, the assay turn-around-time (TAT) from the time of node removal to the report of the assay result to the surgeon. | 1 day
To determine, under clinical use conditions, whether the assay result was or was not received in time ('time for decision' (TFD)) to make an intra-operative decision to proceed to further non-sentinel axillary lymph node dissection. | 1 day
To collect data in relation to other surgical procedures during the SLND/breast surgery to determine if the assay TAT resulted in longer surgery time than would have occurred if the assay had not been used. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Scott U Adams, MS, Study Director — Ortho-Clinical Diagnostics, Inc.
Locations (6):
- United States (6):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - St. Anthony's Hospital, St. Petersburg, Florida
  - Georgia Esoteric and Molecular Labs, LLC, Augusta, Georgia
  - Woman's Hospital, Flowood, Mississippi

REFERENCES:
- [Background] Blumencranz P, Whitworth PW, Deck K, Rosenberg A, Reintgen D, Beitsch P, Chagpar A, Julian T, Saha S, Mamounas E, Giuliano A, Simmons R. Scientific Impact Recognition Award. Sentinel node staging for breast cancer: intraoperative molecular pathology overcomes conventional histologic sampling errors. Am J Surg. 2007 Oct;194(4):426-32. doi: 10.1016/j.amjsurg.2007.07.008. PMID 17826050
- [Background] Veys I, Majjaj S, Salgado R, Noterman D, Schobbens JC, Manouach F, Bourgeois P, Nogaret JM, Larsimont D, Durbecq V. Evaluation of the histological size of the sentinel lymph node metastases using RT-PCR assay: a rapid tool to estimate the risk of non-sentinel lymph node invasion in patients with breast cancer. Breast Cancer Res Treat. 2010 Dec;124(3):599-605. doi: 10.1007/s10549-009-0555-2. Epub 2009 Sep 25. PMID 19779817
- [Background] Julian TB, Blumencranz P, Deck K, Whitworth P, Berry DA, Berry SM, Rosenberg A, Chagpar AB, Reintgen D, Beitsch P, Simmons R, Saha S, Mamounas EP, Giuliano A. Novel intraoperative molecular test for sentinel lymph node metastases in patients with early-stage breast cancer. J Clin Oncol. 2008 Jul 10;26(20):3338-45. doi: 10.1200/JCO.2007.14.0665. PMID 18612150